CLINICAL TRIAL: NCT05138783
Title: Clinical Performance of Two Daily Disposable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-P006
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Refractive Errors
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PRECISION1, then Biotrue (Other): Verofilcon A contact lenses worn first, with nesofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) at least 10 hours per day for 8 -0/+3 days. A fresh pair of lenses will be worn each day.
  Interventions: Device: Verofilcon A contact lenses; Device: Nesofilcon A contact lenses
- Biotrue, then PRECISION1 (Other): Nesofilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) at least 10 hours per day for 8 -0/+3 days. A fresh pair of lenses will be worn each day.
  Interventions: Device: Verofilcon A contact lenses; Device: Nesofilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Spherical soft contact lenses for daily disposable wear
  Other Names: PRECISION1™
Device: Nesofilcon A contact lenses — Spherical soft contact lenses for daily disposable wear
  Other Names: Biotrue® ONEday

SUMMARY:
The purpose of this study is to compare the clinical performance of PRECISION1 contact lenses with Biotrue contact lenses.

DETAILED DESCRIPTION:
Subjects will be expected to attend 3 visits. Subjects will be expected to wear their study contact lenses every day for at least 10 hours per day over an 8-day period for each study lens type. The total duration of a subject's participation in the study will be up to 22 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wear of spherical soft contact lenses with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.
* Willing to wear habitual spectacles for vision correction when study lenses are not worn, as needed.
* Willing to wear contact lenses for at least 16 hours on the day prior to Visit 2 and the day prior to Visit 3.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Participation in a clinical trial within the previous 30 days or currently enrolled in any clinical trial.
* Habitual PRECISION1, Biotrue, and DAILIES TOTAL1 contact lens wear.
* Monovision and multifocal lens wear.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Kindred Optics at Maitland Vision, Maitland, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - Franklin Park Eye Center PC, Franklin Park, Illinois
  - Heart of America Eye Care, Shawnee Mission, Kansas
  - Complete Eye Care Of Medina, Medina, Minnesota
  - ProCare Vision Centers, Inc., Granville, Ohio
  - Clarke EyeCare Center, Wichita Falls, Texas
  - Stine Eye Center, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 8 investigative sites in the US.
Pre-assignment Details: Of the 129 enrolled, 3 subjects were screen failures prior to randomization. This reporting group includes all randomized subjects, as treated (126).
Units Other Than Participants: eyes
Groups:
- PRECISION1, Then Biotrue: Verofilcon A contact lenses worn first, with nesofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) at least 10 hours per day for 8 -0/+3 days. A fresh pair of lenses was worn each day.
- Biotrue, Then PRECISION1: Nesofilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) at least 10 hours per day for 8 -0/+3 days. A fresh pair of lenses was worn each day.
Period: First Wear Period, 8 -0/+3 Days
Arm/Group | PRECISION1, Then Biotrue | Biotrue, Then PRECISION1
Started | 62; 124 eyes | 64; 128 eyes
Completed | 62; 124 eyes | 64; 128 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Second Wear Period, 8 -0/+3 Days
Arm/Group | PRECISION1, Then Biotrue | Biotrue, Then PRECISION1
Started | 62; 124 eyes | 64; 128 eyes
Completed | 62; 124 eyes | 64; 128 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study, as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRECISION1, Then Biotrue | Biotrue, Then PRECISION1 | Total
Number analyzed (Participants) | 62 | 64 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.2) | 33.5 (7.3) | 32.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 20 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 52 | 58 | 110
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57 | 61 | 118
  Black or African American | 2 | 0 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 2 | 1 | 3
  Multi-racial | 0 | 1 | 1
  Missing data | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance Visual Acuity (VA) With Study Lenses
Description: Visual Acuity (VA) was collected for each eye individually with study lenses in place using a letter chart. VA was measured in logarithm of the minimum angle of resolution (logMAR). A logMAR value of 0 corresponds to 20/20 Snellen acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity.
Time Frame: Day 8 (-0/+3 days), each study lens type
Population: Full Analysis Set: All randomized subjects who were exposed to any study lenses evaluated in this clinical study with data at Day 8.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- PRECISION1: Verofilcon A contact lenses worn in Period 1 or Period 2, as randomized, in both eyes during waking hours only at least 10 hours per day for -0/+3 days. A fresh pair of lenses was worn each day.
- Biotrue: Nesofilcon A contact lenses worn in Period 1 or Period 2, as randomized, in both eyes during waking hours only at least 10 hours per day for -0/+3 days. A fresh pair of lenses was worn each day.
Arm/Group | PRECISION1 | Biotrue
Number analyzed (Participants) | 126 | 126
Number analyzed (eyes) | 252 | 252
logMAR | -0.13 (0.006) | -0.13 (0.006)
Statistical Analysis 1: Comparison: PRECISION1 vs Biotrue; Test type: Non-Inferiority — Noninferiority in distance VA was declared if upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least squares mean difference = -0.01, 95% CI 1-sided [upper limit 0.00], Standard Error of Mean 0.004 — LSM results based on mixed effects repeated measures model with both fixed (lens, period, and sequence) and random (subject) effects. Difference = PRECISION1 minus BIOTRUE. Sign (either negative or positive) is retained with the rounded value

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit, up to 22 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses, as treated.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- PRECISION1 Ocular; PRECISION1 NonOcular: Events reported in this group occurred while exposed to the verofilcon A contact lenses.
- Biotrue Ocular; Biotrue NonOcular: Events reported in this group occurred while exposed to the nesofilcon A contact lenses.
Arm/Group | Pretreatment | PRECISION1 Ocular | PRECISION1 NonOcular | Biotrue Ocular | Biotrue NonOcular
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/252 | 0/126 | 0/252 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/252 | 0/126 | 0/252 | 0/126
Other Adverse Events (participants affected / at risk) | 0/126 | 0/252 | 0/126 | 0/252 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study,

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT05138783/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT05138783/SAP_001.pdf